CLINICAL TRIAL: NCT07193030
Title: Peer-Led Intervention To Reduce Alcohol Binge Drinking Among University Students In Romania- A Pilot Study Of The Implementation Processes
Brief Title: Peer-Led Intervention To Reduce Alcohol Binge Drinking Among University Students In Romania
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Rubana Islam, Scientist, International Agency for Research on Cancer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PP202207-30
Record Dates: First submitted 2025-09-04; First posted 2025-09-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Binge Alcohol Consumption; Binge Drinking
Keywords: Binge drinking; Alcohol Brief Intervention; Behaviour change wheel; University students; Romania
MeSH Terms: conditions — Binge Drinking | interventions — Ethanol; Crisis Intervention; Counseling

STUDY DESIGN:
Intervention Model Description: Parallel group cluster randomised trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer led- alcohol brief intervention (Experimental): The intervention arm will receive the brief advice from their peers about binge drinking. The intervention will last 15-20 minutes.
  Interventions: Behavioral: Peer-led Alcohol Brief Intervention (identification + advice)
- No intervention (No Intervention): The control arm will receive no intervention. They will only complete the surveys at three time points.

INTERVENTIONS:
Behavioral: Peer-led Alcohol Brief Intervention (identification + advice) — The intervention consists of a peer-led ABI for university students. This intervention aligns with the ABI approach recommended by the WHO as a cost-effective strategy to reduce harmful alcohol use, particularly in primary care and community settings. The brief advice component of the intervention will incorporate Motivational Interviewing (MI) techniques, a client-centred, evidence-based counselling style intervention effective for reducing risky drinking behaviours. The brief advice will be tailored based on behavioural insights identified through formative research, such as individual perceived facilitators and barriers.
  The Alcohol Use Disorders Identification Test- Consumption (AUDIT-C) will be used as the screening tool for identification.
  A one-on-one Brief Advice sessions of 15-20 minutes will be delivered by trained peer educators, i.e., university students who are not healthcare professionals but have been specifically trained in delivering brief advice.
  Arms: Peer led- alcohol brief intervention

SUMMARY:
The goal of this clinical trial is to learn if a behavioural intervention to change binge drinking habits in university students in Romania is feasible. The main research question is:

Is a peer-led Alcohol Brief Intervention feasible to be implemented in a Romanian University to reduce binge drinking among students?

Researchers will compare brief intervention (counselling) to no intervention.

Student participants will:

1. Receive brief counselling for 15-20 minutes by their peers who were trained.
2. Report their alcohol consumption levels in three surveys conducted over three months.

DETAILED DESCRIPTION:
Pre-intervention focus group discussions: Students will be involved in group discussions, up to 90 minutes, to share their perspective on binge drinking.

Pre-intervention co-design workshop: Students will be involved in a 3-hour workshop to co-design messages to be used during the brief advice intervention.

University staff will be invited to participate in in-depth interviews lasting up to 60 minutes.

Intervention:

Student participants- They will be administered a pre-intervention survey lasting approximately 60-minutes by research assistants, a 15-20 minutes brief advice/counselling session by their peers, a midline survey of 5 minutes, and an endline survey of approximately 60 minutes administered by research assistants. these students will be invited to take part in a focus group at the end of the intervention lasting 90 minutes.

Peers- Peers are students who volunteered to deliver the brief counselling to other students. They will first undergo training by motivational interviewing experts for approximately 6-8 hours spread across 2 days. We intend to recruit 4 peers and each one will deliver the brief advice to 15 students, each session lasting 15-20 minutes. The peers will then be invited to participate in a focus group discussion lasting up to 90 minutes at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* University students currently enrolled in full-time undergraduate or postgraduate programs at Babeș-Bolyai University in Romania
* Able to provide informed consent
* Willing to participate in an in-person session
* Alcohol status: AUDIT-C scoring 3 or above in females, 4 or above in males

Exclusion Criteria:

* Students currently receiving treatment for alcohol dependence or any other substance use disorder
* Students with a diagnosed severe mental health condition that may impair participation
* Participation in any similar alcohol reduction program in the past 6 months.
* Abstinent from alcohol consumption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline, 3 month
  Number of participants recruited
Retention rate | Baseline, 3 month
  Number of participants retained
Knowledge on binge drinking and adverse outcomes | Baseline, 1 month, 3 month
  Change in knowledge on binge drinking and adverse outcomes. Ad hoc questions developed for this study will be used. Scoring will be done on the number questions answered correctly.
Attitude | Baseline, 3 month
  Change in attitude to binge drinking using the Theory of Planned Behaviour tool (by Cooke, R., 2007). A 7-point Likert scale will be used on five bipolar scales (harmful-beneficial, unpleasant-pleasant, bad-good, worthless-valuable, unenjoyable-enjoyable.
Subjective norms | Baseline, 3 month
  Change in subjective norms using the Theory of Planned Behaviour tool. A 7 point Likert scale will be used.
Intention to change | Baseline, 3 month
  Change in intention change using the Theory of Planned Behaviour tool. A 7 point Likert scale will be used.
Feasibility outcome | end line (month 3)
  This will be explored qualitatively asking questions about study acceptability, appropriateness, and fidelity using semi-structured interview guidelines. (Note: This is a qualitative outcome; no scoring will be done)

SECONDARY OUTCOMES:
Change in frequency of binge drinking in the past four weeks | Baseline, 1 month, 3month
  measured via self-report using AUDIT-C, e.g. number of binge episodes, ≥6 drinks or 60 g of pure alcohol on one occasion

CONTACTS AND LOCATIONS:
Overall Officials: Rubana Islam, PhD, Principal Investigator — IARC; Carolina Espina, PhD, Study Director — IARC

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because of confidentiality concerns and the sensitive nature of the information collected. The trial was not designed with participant consent for public data sharing, and de-identification would not fully eliminate the risk of re-identification. Findings will instead be disseminated through aggregated results in publications and reports.

REFERENCES:
- [Background] DeBerardinis RJ, Kazazian HH Jr. Analysis of the promoter from an expanding mouse retrotransposon subfamily. Genomics. 1999 Mar 15;56(3):317-23. doi: 10.1006/geno.1998.5729. PMID 10087199
- [Background] Glanz K, Bishop DB. The role of behavioral science theory in development and implementation of public health interventions. Annu Rev Public Health. 2010;31:399-418. doi: 10.1146/annurev.publhealth.012809.103604. PMID 20070207
- [Background] Mirowski M, Atlas P. [Importance of the precordial derivations for the diagnosis of auricular rhythms]. Arch Mal Coeur Vaiss. 1970 Feb;63(2):190-8. No abstract available. French. PMID 4985973